CLINICAL TRIAL: NCT04706767
Title: Effects of Lidocaine, Dexmedetomidine, and Their Combination on Quality of Recovery Undergoing Laparoscopic Total Hysterectomy
Brief Title: Effect of Co-administration Lidocaine and Dexmedetomidine on Quality of Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anqing Municipal Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: xuzhang
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Lidocaine; Dexmedetomidine; Quality of Recovery(QoR-40), Preoperative and Postoperative
Keywords: Lidocaine; Dexmedetomidine; Quality of recovery
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Effect of Co-administration Lidocaine and Dexmedetomidine on Quality of Recovery (Experimental)
  Interventions: Drug: Co-administration Lidocaine and Dexmedetomidine; Drug: Dexmedetomidine infusion; Drug: Lidocaine infusion; Drug: Saline infusion
- Effect of Dexmedetomidine infusion on Quality of Recovery (Experimental)
  Interventions: Drug: Co-administration Lidocaine and Dexmedetomidine; Drug: Dexmedetomidine infusion; Drug: Lidocaine infusion; Drug: Saline infusion
- Effect of Lidocaine infusion on Quality of Recovery (Experimental)
  Interventions: Drug: Co-administration Lidocaine and Dexmedetomidine; Drug: Dexmedetomidine infusion; Drug: Lidocaine infusion; Drug: Saline infusion
- Effect of saline infusion on Quality of Recovery (Experimental)
  Interventions: Drug: Co-administration Lidocaine and Dexmedetomidine; Drug: Dexmedetomidine infusion; Drug: Lidocaine infusion; Drug: Saline infusion

INTERVENTIONS:
Drug: Co-administration Lidocaine and Dexmedetomidine — Patients received a bolus infusion of lidocaine (2%; 1.5 mg/kg) and dexmedetomidine (0.5 µg/kg) over 10 min before the induction of anesthesia, and then lidocaine and dexmedetomidine were infused at a rate of 1.5 mg/kg/h and 0.4 µg/kg/h until close of the pneumoperitoneum, respectively.
Drug: Dexmedetomidine infusion — Patients received a bolus infusion of dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until close of the pneumoperitoneum.
Drug: Lidocaine infusion — Patients received a bolus infusion of lidocaine (2%; 1.5 mg/kg over 10 min before the induction of anesthesia), and then lidocaine was infused at a rate of 1.5 mg/kg/h until close of the pneumoperitoneum.
Drug: Saline infusion — Patients received the same volume of normal saline 10 min before the induction of anesthesia, and then normal saline (0.9%) was continuously infused in an equal volume until close of the pneumoperitoneum.

SUMMARY:
BACKGROUND: Some studies have revealed that intravenous (IV) lidocaine or dexmedetomidine might improve the quality of recovery undergoing laparoscopic surgery. The investigators investigated whether co-administration lidocaine and dexmedetomidine could better improve the the quality of recovery after laparoscopic total hysterectomy.

METHODS: One hundred and forty-four women with elective laparoscopic total hysterectomy were randomly divided into four groups: Patients in group L received a bolus infusion of lidocaine (2%; 1.5 mg/kg over 10 min before the induction of anesthesia), and then lidocaine was infused at a rate of 1.5 mg/kg/h until close the pneumoperitoneum. Patients in group D received a bolus infusion of dexmedetomidine (0.5 µg/kg over 10 min before the induction of anesthesia), and then dexmedetomidine was infused at a rate of 0.4 μg/kg/h until close the pneumoperitoneum. Patients in group LD received a bolus infusion of lidocaine (2%; 1.5 mg/kg) and dexmedetomidine (0.5 µg/kg) over 10 min before the induction of anesthesia, and then lidocaine and dexmedetomidine were infused at a rate of 1.5 mg/kg/h and 0.4 µg/kg/h until close the pneumoperitoneum, respectively. Patients in group C received the same volume of normal saline 10 min before the induction of anesthesia, and then normal saline (0.9%) was continuously infused in an equal volume until close the pneumoperitoneum. Primary outcome was the quality of recovery (QoR-40) at 1 day prior to sugery, 1 day after sugery, and 2 days after sugery. The secondary outcomes included perioperative remifentanil consumption, postoperative VAS scores, the incidence of postoperative nausea and vomiting, postoperative rescue analgesics and anti-emetics, recovery time, extubation time, and Ramsay sedation scale at 5 min, 10min, 30 min, 60 min after extubation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical statusⅠand Ⅱ
* Scheduled for elective laparoscopic total hysterectomy

Exclusion Criteria:

* History of allergy to local anesthetics
* BMI>30
* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative opioids medication and psychiatric
* preoperative bradycardia
* preoperative atrioventricular block

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Quality of recovery scores(QoR-40) | 1 day after operation
  Our primary outcome was Quality of recovery scores(QoR-40) 1 day after operation

SECONDARY OUTCOMES:
Intraoperative remifentanil total dose | Intraoperative
  Secondary Outcome Measure was remifentanil total dose during the perioperative period
Recovery time | Immediately after the surgery
  Secondary Outcome Measure was recovery time
Extubation time | Immediately after the surgery
  Secondary Outcome Measure was extubation time
Pain visual analogue scale scores | The first 24 hours after operation
  Secondary Outcome Measure was pain visual analogue scale scores
PONV scores | The first 24 hours after operation
  Secondary Outcome Measure was PONV scores
The consumption of sufentanil | The first 24 hours after operation
  Secondary Outcome Measure was consumption of sufentanil
The length of post-anesthesiacare unit stay | Immediately after the surgery
  Secondary Outcome Measure was the length of post-anesthesiacare unit stay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China